CLINICAL TRIAL: NCT00012688
Title: Periodontal Care and Glycemic Control in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Colgate-Periogard-Dentsply (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DII 99-206
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes Mellitus; Poor Glycemic Control; Peridontal Disease
MeSH Terms: conditions — Diabetes Mellitus | interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Doxycycline HCI 10mg po for 2 weeks; Procedure: Ultrasonic scaling with 0.12% chlorhexidine gluconate

INTERVENTIONS:
Drug: Doxycycline HCI 10mg po for 2 weeks
Procedure: Ultrasonic scaling with 0.12% chlorhexidine gluconate

SUMMARY:
Diabetes is a prevalent and costly disease among users of VA care. Goals of diabetes care include the prevention and/or delay of complications via adequate glycemic control. Improvements in periodontal status may also improve diabetes control.

DETAILED DESCRIPTION:
Background:

Diabetes is a prevalent and costly disease among users of VA care. Goals of diabetes care include the prevention and/or delay of complications via adequate glycemic control. Improvements in periodontal status may also improve diabetes control.

Objectives:

This project will determine the efficacy of a program of periodontal screening and therapy in improving the level of glycemic control in poorly controlled diabetics.

Methods:

Status:

Subject accrual is complete. Data collection is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Patients must have diabetes mellitus, and HbAlc >9, >8 teeth, and CPITN scores of 3 or 4 in, at least 2 sextants of the mouth, indicating moderate to high peridontal treatment need.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Jones, DDS DSc MPH, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

REFERENCES:
- [Result] McCoy LC, Wehler CJ, Rich SE, Garcia RI, Miller DR, Jones JA. Adverse events associated with chlorhexidine use: results from the Department of Veterans Affairs Dental Diabetes Study. J Am Dent Assoc. 2008 Feb;139(2):178-83. doi: 10.14219/jada.archive.2008.0134. PMID 18245686
- [Result] Janket SJ, Jones J, Rich S, Miller D, Wehler CJ, Van Dyke TE, Garcia R, Meurman JH. The effects of xerogenic medications on oral mucosa among the Veterans Dental Study participants. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Feb;103(2):223-30. doi: 10.1016/j.tripleo.2006.05.013. Epub 2006 Aug 4. PMID 17234540
- [Result] Jones JA, Miller DR, Wehler CJ, Rich SE, Krall-Kaye EA, McCoy LC, Christiansen CL, Rothendler JA, Garcia RI. Does periodontal care improve glycemic control? The Department of Veterans Affairs Dental Diabetes Study. J Clin Periodontol. 2007 Jan;34(1):46-52. doi: 10.1111/j.1600-051X.2006.01002.x. Epub 2006 Nov 24. PMID 17137468
- [Result] Jones JA, Miller DR, Wehler CJ, Rich S, Krall E, Christiansen CL, Rothendler JA, Garcia RI. Study design, recruitment, and baseline characteristics: the Department of Veterans Affairs Dental Diabetes Study. J Clin Periodontol. 2007 Jan;34(1):40-5. doi: 10.1111/j.1600-051X.2006.00998.x. Epub 2006 Oct 13. PMID 17040483
- [Result] Cunha-Cruz J, Hujoel PP, Kressin NR. Oral health-related quality of life of periodontal patients. J Periodontal Res. 2007 Apr;42(2):169-76. doi: 10.1111/j.1600-0765.2006.00930.x. PMID 17305876